CLINICAL TRIAL: NCT03863587
Title: A Randomized, Parallel-controlled, Intravenous Single-dose, Phase I Clinical Study Comparing the Pharmacokinetic Profile, Safety, Tolerability and Immunogenicity of HLX12 and Cyramza (Ramucirumab) in Healthy Male Adult Subjects
Brief Title: Compare Pharmacokinetic, Safety, Tolerability and Immunogenicity of HLX12 and Ramucirumab in Healthy Male Adult Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated prematurely due to the difficulty in recruiting participants caused by the COVID-19 pandemic.
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HLX12-001
Record Dates: First submitted 2019-02-25; First posted 2019-03-05 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — Ramucirumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX12 group (Experimental): HLX12 are given intravenous infusion 8 mg/kg, prepared with normal saline to an administration volume of 250 mL, and the administration time is 90 min (± 10 min).
  Interventions: Biological: HLX12
- Cyramza (Ramucirumab) group (Active Comparator): Ramucirumab are given intravenous infusion of Cyramza 8 mg/kg, prepared with normal saline to an administration volume of 250 mL, and the administration time is 90 min (± 10 min).
  Interventions: Biological: Cyramza (Ramucirumab)

INTERVENTIONS:
Biological: HLX12 — healthy volunters receive HLX12 (8mg/kg) once
  Arms: HLX12 group
Biological: Cyramza (Ramucirumab) — healthy volunters receive Cyramza (Ramucirumab) 8mg/kg once
  Arms: Cyramza (Ramucirumab) group

SUMMARY:
The study consists of 2 parts:

Part I study: to preliminarily compare the PK profile of HLX12 and Cyramza This study is an open-label, randomized, parallel-controlled, intravenous single-dose pretrial study comparing the pharmacokinetic profile, safety, tolerability and immunogenicity of HLX12 and Ramucirumab in healthy male adult subjects. The number of subjects is set to 24, who will be randomized into two groups, and each group has the same number of subjects (n=12). Group 1 will receive intravenous infusion of the test preparation T HLX12, while Group 2 will receive Cyramza, once in both groups.

Part II study: to compare the PK similarity between HLX12 and Cyramza This study is a randomized, double-blind, parallel-controlled, intravenous single-dose Phase I clinical study comparing the pharmacokinetic profile, safety, tolerability and immunogenicity of HLX12 and Ramucirumab in healthy male adult subjects.The number of subjects is set to 128, and the treatment is the same with Part I study.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult male aged 18-50 years (including 18 and 50 years old) with a body mass index of 18-28 kg/m2 (including 18 kg/m2 and 28 kg/m2), weighing ≥50 kg and ≤80 kg;

Exclusion Criteria:

Previous or current atopic allergies, hypersensitivity reactions, or allergic reactions that are clinically significant, including known or suspected clinically relevant drug allergies to a component of the study drug or the control drug; Any disease that may affect the safety of the subject or affect the study operation and assessment, according to the investigator's judgment; Have undergone surgery in the past 8 weeks, or are planned for surgery during the study period; Have been inoculated with live virus vaccine within 4 weeks prior to screening, or intend to be inoculated with live virus vaccine during the study period until the end of the last follow-up; Any prior history of exposure to anti-VEGF or anti-VEGF receptor monoclonal antibodies/proteins; Exposure to any monoclonal antibody within 12 months prior to study drug administration; Have used any clinical study drug within 3 months prior to screening, or are still in the follow-up period of a clinical study; Have taken non-steroidal anti-inflammatory drugs (NSAIDs) within 14 days prior to the study drug administration, including any dose of aspirin. NSAIDs (except acetaminophen) shall not be used during the study; QTc interval > 450 ms; ECG is abnormal and the abnormality is clinicaly significant as judged by the investigator; Have taken any alcoholic products within 48 hours prior to the study drug administration; Subjects who have a family history of hypertension, or are found with abnormal blood pressure at screening or on admission to the study site (Day-1): systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, which is judged by the investigator as clinically significant ; Have a genetic predisposition to bleeding or thrombosis, or a history of bleeding due to non-trauma (ie, bleeding requiring medical intervention), a thromboembolic event, or any condition that may increase the risk of bleeding, including coagulopathy, thrombocytopenia (platelet count <100*109/L) or international normalized ratio (INR) higher than 1.5;

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
AUC0~inf | from predose to 1680 hours (Day 71),18 timepoints
  Area under curve from zero to infinity

SECONDARY OUTCOMES:
safety and tolerability of two groups | from day1 to day 71
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
safety and tolerability of two groups | from day1 to day 71
  Number of AE as assessed by CTCAE v5.0
safety and tolerability of two groups | from day1 to day 71
  AE listing as assessed by CTCAE v5.0
AUC0~t | from predose to 1680 hours (Day 71),18 timepoints
  area under the concentration-time curve
Cmax | from predose to 1680 hours (Day 71),18 timepoints
  maximum concentration

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Principal Investigator — First Hospital of Jinlin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Background] American Society for Clinical Pharmacology and Therapeutics. Clin Pharmacol Ther. 2022 Mar;111 Suppl 1:S5-S80. doi: 10.1002/cpt.2521. No abstract available. PMID 35132630